CLINICAL TRIAL: NCT06045624
Title: A Phase 1, First in Human, Double-Blind, Placebo-Controlled, Single and Multiple Ascending Dose and Open Label Food Effect Study to Evaluate Safety, Tolerability, and Pharmacokinetics of OR-101 Administered Orally in Healthy Subjects
Brief Title: A First in Human Single and Multiple Ascending Dose and Open Label Food Effect Study of OR-101 in Healthy Subjects
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: The study was cancelled as the sponsor decided to reformulate the IP
Sponsor: Ornovi, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: OR101-HS101
Record Dates: First submitted 2023-09-13; First posted 2023-09-21 (Actual); Last update posted 2024-04-05 (Actual); Status verified 2024-04

CONDITIONS: Alopecia Areata
MeSH Terms: conditions — Alopecia Areata

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Part A (Experimental): Drug- OR-101
  Dosage level: SAD participants will receive either placebo or one of planned doses levels of 15mg, 45mg, 150mg, 450mg, 900mg, 1500mg OR-101 in dose escalating manner in cohorts 1-6.
  Dosage form: Solution
  Route of administration- Oral
  Interventions: Drug: OR-101 (Single ascending dose)
- Part B (Experimental): Drug- OR101
  Dosage level: Food effect participants (8 subjects in 9 cohorts) will only receive OR-101with a high fat meal prior to administration and subjects in corresponding dose under fasted condition will serve as their reference group.
  Dosage form: Solution
  Route of administration- Oral
  Interventions: Drug: OR-101 (Food effect)
- Part C (Experimental): Drug- OR-101
  Dosage level: MAD participants will receive either placebo or one of planned doses levels of 15mg, 45mg, 135mg, 270mg, 540mg and 900mg OR-101 in dose escalating manner in cohorts 1-6. Total dosage of cohort 7 and 8 will be decided based on Safety review committe's input where cohort 8 will receive this daily for 7 days.
  Dosage form: Solution
  Route of administration- Oral
  Interventions: Drug: OR-101 (Multiple ascending dose)
- Placebo (Placebo Comparator): Placebo comparators taken by participants randomised to the placebo arm across Part A and C of the study.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: OR-101 (Single ascending dose) — SAD participants will receive either placebo or one of planned doses levels of 15mg, 45mg, 150mg, 450mg, 900mg, 1500mg OR-101 in dose escalating manner in cohorts 1-6.
  Arms: Part A
Drug: OR-101 (Food effect) — Food effect participants (8 subjects in 9 cohorts) will only receive OR-101with a high fat meal prior to administration and subjects in corresponding dose under fasted condition will serve as their reference group
  Arms: Part B
Drug: OR-101 (Multiple ascending dose) — MAD participants will receive either placebo or one of planned doses levels of 15mg, 45mg, 135mg, 270mg, 540mg and 900mg OR-101 in dose escalating manner in cohorts 1-6. Total dosage of cohort 7 and 8 will be decided based on Safety review committe's input where cohort 8 will receive this daily for 7 days
  Arms: Part C
Drug: Placebo — Participants will receive matching placebo across Part A and C of the study
  Arms: Placebo

SUMMARY:
This first in human phase 1 study to Study will evaluate safety, tolerability, and pharmacokinetics of Single Ascending dose (SAD), Food effect (FE) and Multiple ascending dose (MAD) of OR-101 Administered Orally in healthy subjects

DETAILED DESCRIPTION:
There are three phases of the study: Single ascending dose (SAD), food effect (FE), and multiple ascending dose (MAD) phases.

In the SAD and MAD Phases, up to 64 subjects in each phase may be enrolled in the study. Fortyeight subjects will be randomised in the initial six cohorts; upto 16 subjects may be enrolled in two additional cohorts. For each dose cohort a total of 8 subjects (6 receiving OR-101 and 2 placebo) will be enrolled and randomized.

In the FE phase, up to 8 subjects who will receive a high fat meal prior to administration of OR101 may be enrolled in the study. Subjects who discontinue prior to completion may be replaced at the discretion of the Sponsor and the Investigator.

The SRC including the Investigator, Medical Monitor, Study Director as well as other ad hoc representatives as appropriate will regularly monitor all aspects of subject safety throughout this study. The SRC will review all available, cumulative safety and PK data in a blinded manner to assess the safety of each dose level of OR-101 prior to escalating to the next dose level.

ELIGIBILITY:
Inclusion Criteria:

1. Is willing to sign and date IRB-approved ICF.
2. Is a man or woman between the ages of 18 and 55, inclusive.
3. Has a BMI of 18.0 to 30.5 kg/m2 and a total body weight >50 kg for a man and >45 kg for a woman at Screening and Check-in of Day -1.
4. Is in good health as determined by medical history, PE, clinical laboratory studies, ECGs, VS, and Investigator's judgement (repeat tests are allowed at PI's discretion).
5. Is willing to minimize sun exposure, avoid phototherapy, and not to use tanning beds, tanning booths, or sun lamps during the study (Day 1 to EOS).
6. If a woman of childbearing potential, must not be pregnant, lactating, or planning to become pregnant during the study.
7. Willing to follow the methods of contraception as per the protocol.

Exclusion Criteria:

1. Has any condition that precludes a subject's ability to comply with study requirements, including completion of the study visits.
2. Has a history or current evidence of a clinically significant cardiovascular, respiratory, endocrine, gastrointestinal, renal, hepatic, hematologic, immunologic, genitourinary, dermatological, psychiatric or neurologic abnormality or disease or other medical disorder, including cancer or malignancies.
3. Has clinically significant abnormal laboratory test values as determined by the Investigator or the local or Sponsor Medical Monitor.
4. has BP and HR measurement after 5 minutes rest in a supine position of:

   * systolic BP >150 or <90 mmHg
   * diastolic BP of >95 or <45 mmHg
   * HR >100 or <50 bpm
   * 2 repeats of the subject's BP or HR are permitted for eligibility purposes
5. Has a history of, or currently has, any clinically significant ECG finding, or a QT interval corrected by Fridericia's method (QTcF) of > 450 msec for males and > 470 msec for females.
6. Has unacceptable COVID-19 test results (if required per site policy at the time of enrollment).
7. Has a history of HIV, or hepatitis B or C, or positive serology. Note: Subjects with a history of hepatitis C who have been treated and cured (no detectable HCV RNA) are allowed.
8. Has a history of tuberculosis.
9. Has an active immune suppressed condition or disease.
10. Has a history of recurrent HSV infections (HSV 1 and/or 2) requiring chronic antiviral suppressive therapies (defined as greater than 4 episodes or breakout per calendar year).
11. Is unable to swallow study drug or has a known intolerance or hypersensitivity to OR-101 or any of the excipients contained in the study drug.
12. Has participated in a clinical study and received active treatment during the last 30 days or 5 half-lives, whichever is longer, prior to Day 1.
13. Has received any prescription medication within the last 14 days prior to Day 1 or nonprescription OTC medication within the last 7 days prior to Day 1, or supplement (e.g., St John's wort, echinacea, kava kava, and common valerian) that may induce/inhibit CYP isozymes within the last 30 days or 5 half-lives, whichever is longer, prior to Day 1.

    Note: acetaminophen (paracetamol) or ibuprofen are permitted medications on an as needed basis.
14. Has recent history (within 6 months of screening) of alcohol or drug abuse.
15. Consumes more than 14 units of alcohol per week (7 days) for at last 30 days prior to Day 1 and throughout the end of the study or those who have a history of alcohol or drug/chemical abuse Note: 1 unit of alcohol is equivalent to 240 mL of beer, 120 mL of wine, or 30 mL of spirits.
16. Consumes greater than 500 mg of caffeine or xanthine-containing products per day (e.g., approximately five 240-mL cups of coffee, ten 240-mL cups of tea, twelve 360-mL cans of soft drinks, energy drinks) for at last 30 days prior to Day 1 and throughout the end of the study.
17. Is an active smoker and/or has used nicotine or nicotine-containing products (e.g., nicotine patch and electronic cigarette) within 3 months of Day 1 (to be confirmed by carbon monoxide breath test).
18. Refuses to abstain from alcohol, grapefruit, or Seville-orange containing foods (e.g., orange marmalade) or beverages, from 48 hours prior to Day 1 through the end of the study.
19. Has donated blood > 500 mL within 60 days prior to the Screening Visit (Plasma donation is allowed).
20. Is an employee of Ornovi Pty Ltd or the CRO, or has an immediate family member who is an employee of Ornovi Pty Ltd or the CRO.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2023-10-17 (Estimated); Primary Completion 2024-02-06 (Actual); Study Completion 2024-02-06 (Actual)

PRIMARY OUTCOMES:
Number of participants with Treatment emergent Adverse events (TEAEs) | Upto 8 days in SAD and FE Phase; Upto 14 days in MAD Phase
Number of participants with Serious Adverse events (SAEs) | Upto 8 days in SAD and FE Phase; Upto 14 days in MAD Phase
Number of participants with changes in 12-lead ECG findings | Upto 8 days in SAD and FE Phase; Upto 14 days in MAD Phase
Number of participants in clinical laboratory tests | Upto 8 days in SAD and FE Phase; Upto 14 days in MAD Phase

SECONDARY OUTCOMES:
PK Parameters: Maximum Concentration (Cmax) | SAD and FE- Day1, Day2, Day 3, Day 4 and day 8 post dose; MAD- Day 1 to Day 14 post dose
PK Parameters: Tmax | SAD and FE- Day1, Day2, Day 3, Day 4 and day 8 post dose; MAD- Day 1 to Day 14 post dose
PK Parameters: Area under the curve (AUC) | SAD and FE- Day1, Day2, Day 3, Day 4 and day 8 post dose; MAD- Day 1 to Day 14 post dose
PK Parameters: half life (t1/2) | SAD and FE- Day1, Day2, Day 3, Day 4 and day 8 post dose; MAD- Day 1 to Day 14 post dose
Urine PK Parameters: Renal Clearance (CLr) | SAD Phase only: Urine PK samples at predose void on Day 1, and at 0-4, 4-8, 8-12, 12-24, 24-36, 36-48, 48-60, 60-72 hours postdose.
Urine PK Parameters: nonrenal Clearance (CLnr) | SAD Phase only: Urine PK samples at predose void on Day 1, and at 0-4, 4-8, 8-12, 12-24, 24-36, 36-48, 48-60, 60-72 hours postdose.

CONTACTS AND LOCATIONS:
Locations (1):
- SCIENTIA Clinical Research Ltd, Randwick, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: No